CLINICAL TRIAL: NCT02577822
Title: The Viability of Short Stems in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, David W. Manning, Associate Professor, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STU00082654
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis of Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Short Stem Group (Other): Short femoral stem
  Interventions: Device: Taperloc short length stem
- Long Stem Group (Other): standard-length stem
  Interventions: Device: Taperloc standard length stem

INTERVENTIONS:
Device: Taperloc standard length stem
  Arms: Long Stem Group
Device: Taperloc short length stem
  Arms: Short Stem Group

SUMMARY:
The purpose of this study is to determine the viability of short femoral stems as an alternative to standard-length stems in total hip arthroplasty.

DETAILED DESCRIPTION:
Porous-coated cementless stems were introduced in the late 1970s, in response to the high incidence of aseptic loosening associated with cemented stems (Judet et al 1978, Kavanagh et al 1989, Lord 1982, Stauffer 1982). The stem's porous surface achieves fixation via bony ingrowth at the endosteum (Engh et al 1987). In an effort to mimic the femur's natural stress distribution, many designs preferentially load the metaphysis (Joshi et al 2000). One such design is the proximally coated titanium tapered wedge, which is widely used today (Pitto et al 2010). Because loading is primarily dictated by bony ingrowth, the proximal porous coating avoids fixation at the diaphysis. The flat, tapered geometry reduces stiffness compared to cylindrical stems, thereby propagating stress to the proximal femur, rather than down the stem's axis (Engh et al 1987, Harvey et al 1999), (Boehm 1998). Further contributing to decreased stiffness is titanium's low elastic modulus, relative to that of cobalt-chromium (Harvey et al 1999, Mulliken et al 1996). Some contend the need for distal fixation in Dorr type C hips due to thin cortical bone at the metaphysis; however, proximally engaging stems have been shown to perform well in these patients (Kelly et al 2007, Reitman et al 2003).

If a stem's objective is to load proximally, then perhaps it need not extend into the diaphyseal canal. The emergence of short stems has initiated an alternative means of proximal loading, without the disruption of diaphyseal bone stock. The smaller incisions involved with short stem total hip arthroplasty (THA) reduce damage to muscle and soft tissue (Molli et al 2012). This enables a faster, more complete recovery for the patient, as well as a cosmetically superior result (Sherry et al 2003). Additionally, the preservation of bioavailable bone can be advantageous if a revision surgery is required (Toth et al 2010). Because short stems do not extend into the diaphysis, issues regarding proximal-distal mismatch of the femur are avoided (Patel et al 2013). This eases implantation and reduces the risk of intraoperative fracture (Azzam et al 2010, Cooper & Rodriguez 2010). The risk of intraoperative fracture is further mitigated because short stem THA does not require the use of reamers (Molli et al 2012, Scott et al 1975, Taylor et al 1978).

Although the standard-length proximally coated titanium tapered wedge has a successful long-term track record, its design leaves room for improvement (Mallory et al 2001, Marshall et al 2004). Standard length stems cause stress-shielding in Gruen zones 1 and 7, suggesting that the diaphyseal portion of a stem may interfere with proximal loading (Gibbons et al 2001, Schmidt et al 2004). Even proximally coated flat tapered stems are subject to diaphyseal loading (Cooper et al 2011). The Accolade stem has been associated with significant early subsidence, especially in males with Dorr type A hips (Jacobs & Christensen 2009). This suggests that the stem may wedge distally, thereby interfering with osseointegration (White et al 2012). By achieving a purely metaphyseal fit, short stems can prevent excessive bone loss secondary to stress shielding (Gustke 2012). The investigators believe short stems are an equally effective alternative to traditional tapered stems in THA; however, long-term studies are essential to proving their efficacy.

Long-term studies of short stems are lacking in current literature. With respect to initial stability and bony ingrowth, short-term data is promising; however, there is still potential for late aseptic failure (Capello et al 2009, Kroell et al 2009, Morales de Cano et al 2013, Schmidutz et al 2012). By conducting a single blinded, prospective, randomized investigation of two stems of varying length with equal metallurgy, coating, and proximal geometry, the investigators can identify the effects of stem length on long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Must require a total hip arthroplasty.
* Ages 18-85 years, regardless of gender, ethnicity, or pathology

Exclusion Criteria:

* This study excludes any populations at risk.
* Minors, as well as any persons unable to consent, will not be eligible.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Department of Orthopaedic Surgery, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Stem Group: Short femoral stem
  Taperloc short length stem
- Long Stem Group: standard-length stem
  Taperloc standard length stem
Period: Overall Study
Arm/Group | Short Stem Group | Long Stem Group
Started | 27 | 33
Completed | 21 | 20
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Stem Group | Long Stem Group | Total
Number analyzed (Participants) | 27 | 33 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.28 (10.73) | 58.70 (11.99) | 60.47 (11.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 17 | 32
  Male | 12 | 16 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 14 | 16 | 30
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 27 | 33 | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean VR-12 Mental Composite Score Through 2 Years Post Operative
Description: Veteran's RAND 12 Item Health Survey used to assess health-related quality of life, to estimate disease burden, and to evaluate disease-specific benchmarks. Scores for the Mental Composite Score (MCS) range from 5.2 to 76.3 and are evaluated as a summative T-score with population mean of 50 (Standard Deviation = 10);higher scores indicate improved mental wellness/function as reported by patients.
Time Frame: Assesed pre-operatively, 6 weeks post-operatively, 3 months post-operatively, 6 months post-operatively, 12 months post-operatively, and 2 years post-operatively.
Population: Discrepancies between the total number of patients analyzed and patients included in participant flow is due to patients lost to follow-up during the course of the study despite attempts to contact them by the research team
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 27 | 33
T-Score
  VR-12 MCS Mean Score (Pre-Op): number analyzed (Participants) | 26 | 30
  VR-12 MCS Mean Score (Pre-Op) | 47.3 (11.3) | 50.6 (13.8)
  VR-12 MCS Mean Score (6 wk): number analyzed (Participants) | 24 | 28
  VR-12 MCS Mean Score (6 wk) | 54.9 (8.9) | 53.8 (11.7)
  VR-12 MCS Mean Score (3 mo): number analyzed (Participants) | 27 | 27
  VR-12 MCS Mean Score (3 mo) | 56.4 (11.2) | 56.9 (10.6)
  VR-12 MCS Mean Score (6 mo): number analyzed (Participants) | 25 | 30
  VR-12 MCS Mean Score (6 mo) | 54.8 (10.2) | 56.4 (9.3)
  VR-12 MCS Mean Score (1 yr): number analyzed (Participants) | 23 | 27
  VR-12 MCS Mean Score (1 yr) | 53.0 (9.6) | 56.7 (8.3)
  VR-12 MCS Mean Score (2 yr): number analyzed (Participants) | 14 | 12
  VR-12 MCS Mean Score (2 yr) | 52.3 (9.9) | 55.3 (9.9)

2. Primary Outcome: Mean VR-12 Physical Composite Score Through 2 Years Post Operative
Description: Veteran's RAND 12 Item Health Survey used to assess health-related quality of life, to estimate disease burden, and to evaluate disease-specific benchmarks. Scores for the Physical Composite Score (PCS) range from 6.3 to 71.8 and are evaluated as a summative T-score with population mean of 50 (Standard Deviation = 10);higher scores indicate improved mental wellness/function as reported by patients.
Time Frame: Assessed pre-operatively, 6 weeks post-operatively, 3 months post-operatively, 6 months post-operatively, 12 months post-operatively, and 2 years post-operatively.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 27 | 33
T-Score
  VR-12 PCS Mean Score (Pre-Op): number analyzed (Participants) | 26 | 30
  VR-12 PCS Mean Score (Pre-Op) | 25.2 (6.8) | 23.6 (5.3)
  VR-12 PCS Mean Score (6 wk): number analyzed (Participants) | 24 | 28
  VR-12 PCS Mean Score (6 wk) | 37.0 (10.0) | 37.8 (9.8)
  VR-12 PCS Mean Score (3 mo): number analyzed (Participants) | 27 | 27
  VR-12 PCS Mean Score (3 mo) | 42.1 (10.2) | 40.1 (10.6)
  VR-12 PCS Mean Score (6 mo): number analyzed (Participants) | 25 | 30
  VR-12 PCS Mean Score (6 mo) | 45.8 (10.0) | 44.7 (9.5)
  VR-12 PCS Mean Score (1 yr): number analyzed (Participants) | 23 | 27
  VR-12 PCS Mean Score (1 yr) | 48.7 (10.9) | 49.5 (8.3)
  VR-12 PCS Mean Score (2 yr): number analyzed (Participants) | 14 | 12
  VR-12 PCS Mean Score (2 yr) | 45.1 (11.3) | 48.5 (5.2)

3. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Pain Behavior Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Pain Behavior domain higher scores indicate more frequent and severe incidence of pain during daily activities
Time Frame: Pre-operatively, 6 weeks post-operatively, 3 months post-operatively, 6 months post-operatively, 12 months post-operatively, and 2 years post-operatively.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 27 | 33
T-Score
  Pain Behavior T-Score (Pre-Op): number analyzed (Participants) | 27 | 30
  Pain Behavior T-Score (Pre-Op) | 59.2 (6.5) | 61.3 (4.2)
  Pain Behavior T-Score (6 wk): number analyzed (Participants) | 27 | 30
  Pain Behavior T-Score (6 wk) | 51.9 (9.1) | 51.0 (10.4)
  Pain Behavior T-Score (3 mo): number analyzed (Participants) | 27 | 30
  Pain Behavior T-Score (3 mo) | 48.0 (10.1) | 52.0 (8.8)
  Pain Behavior T-Score (6 mo): number analyzed (Participants) | 26 | 30
  Pain Behavior T-Score (6 mo) | 47.6 (10.5) | 47.4 (10.8)
  Pain Behavior T-Score (1 yr): number analyzed (Participants) | 26 | 28
  Pain Behavior T-Score (1 yr) | 45.2 (11.0) | 45.2 (9.8)
  Pain Behavior T-Score (2 yr): number analyzed (Participants) | 19 | 19
  Pain Behavior T-Score (2 yr) | 43.8 (10.8) | 40.3 (8.7)

4. Secondary Outcome: EBRA (Ein-Bild-Roentgen-Analyse) Femoral Component Analysis (EBRA-FCA) of Implant Subsidence Through 2 Years Post Operative
Description: EBRA-FCA is a commonly employed technique to evaluate implant migration via radiographic measurements taken over the duration of recovery. The mean subsidence values measured in millimeters were recorded for both the short and standard stem cohorts at each of the clinic visits for SOC.
  Of note, the individual responsible for performing and recording these measurements could not be reached during upload of the final study data and consequently the dispersion values for this measure were not available at the time of publication. The dispersion values for these measures have been recorded as '0' for each time point pending any response from the individual to obtain the original data.
Time Frame: Assessed 6 weeks post-operatively, 6 months post-operatively, 12 months post-operatively, and 2 years post-operatively.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 21 | 20
millimeters
  Femoral Stem Subsidence (6 wk) | 0.124 (0.961) | 0.193 (0.533)
  Femoral Stem Subsidence (6 mo) | 0.448 (1.200) | 0.702 (1.080)
  Femoral Stem Subsidence (1 yr) | 0.526 (1.653) | 1.303 (1.264)
  Femoral Stem Subsidence (2 yr) | 0.590 (1.072) | 1.414 (1.547)

5. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Physical Function Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Physical Function domain higher scores indicated improved physical function as reported by the patient
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 27 | 33
T-Score
  Physical Function T-Score (Pre-Op): number analyzed (Participants) | 27 | 30
  Physical Function T-Score (Pre-Op) | 29.6 (5.8) | 31.7 (6.2)
  Physical Function T-Score (6 wk): number analyzed (Participants) | 27 | 30
  Physical Function T-Score (6 wk) | 41.00 (7.8) | 42.6 (8.00)
  Physical Function T-Score (3 mo): number analyzed (Participants) | 27 | 30
  Physical Function T-Score (3 mo) | 45.5 (8.3) | 45.4 (9.5)
  Physical Function T-Score (6 mo): number analyzed (Participants) | 26 | 30
  Physical Function T-Score (6 mo) | 47.4 (8.6) | 47.9 (8.0)
  Physical Function T-Score (1 yr): number analyzed (Participants) | 26 | 28
  Physical Function T-Score (1 yr) | 48.3 (8.8) | 51.1 (7.1)
  Physical Function T-Score (2 yr): number analyzed (Participants) | 19 | 19
  Physical Function T-Score (2 yr) | 52.9 (12.1) | 53.9 (9.7)

6. Primary Outcome: PROMIS Computerized Adaptive Tests (CATs) for Pain Interference Through 2 Years Post-operative
Description: Patient-reported outcome (PRO) measures use answers that patients provide to questions to produce numeric values which indicate patients' state of wellbeing or suffering as well as their ability or lack of ability to function. Values are reported as T-scores with a reference population mean of 50 (SD=10); for the Pain Interference domain higher scores indicated greater impact on patient's ability to perform daily activities and social function
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Short Stem Group | Long Stem Group
Number analyzed (Participants) | 27 | 33
T-Score
  Pain Interference T-Score (Pre-Op): number analyzed (Participants) | 27 | 30
  Pain Interference T-Score (Pre-Op) | 64.6 (8.6) | 67.4 (6.5)
  Pain Interference T-Score (6 wk): number analyzed (Participants) | 27 | 30
  Pain Interference T-Score (6 wk) | 51.7 (10.3) | 53.1 (9.6)
  Pain Interference T-Score (3 mo): number analyzed (Participants) | 27 | 30
  Pain Interference T-Score (3 mo) | 49.7 (10.1) | 51.1 (10.1)
  Pain Interference T-Score (6 mo): number analyzed (Participants) | 26 | 30
  Pain Interference T-Score (6 mo) | 47.9 (9.8) | 46.6 (10.6)
  Pain Interference T-Score (1 yr): number analyzed (Participants) | 26 | 28
  Pain Interference T-Score (1 yr) | 48.00 (10.5) | 44.0 (8.3)
  Pain Interference T-Score (2 yr): number analyzed (Participants) | 19 | 19
  Pain Interference T-Score (2 yr) | 46.7 (10.5) | 42.2 (6.0)

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored as part of this study
Description: Adverse events were not monitored as part of this study
Arm/Group | Short Stem Group | Long Stem Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT02577822/Prot_SAP_000.pdf
  • Informed Consent Form (2015-08-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT02577822/ICF_001.pdf